CLINICAL TRIAL: NCT02305758
Title: Randomized, Blinded, Multicenter, Phase 2 Study Comparing Veliparib Plus FOLFIRI ± Bevacizumab Versus Placebo Plus FOLFIRI ± Bevacizumab in Previously Untreated Metastatic Colorectal Cancer
Brief Title: Study Comparing Veliparib Plus FOLFIRI Versus Placebo Plus FOLFIRI With or Without Bevacizumab in Previously Untreated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M14-217; 2014-002866-65 (EudraCT Number)
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Untreated Metastatic Colorectal Cancer
Keywords: PARP inhibitor; veliparib; metastatic colorectal cancer; ABT-888; first line; previously untreated; colorectal cancer; colon cancer; rectal cancer; FOLFIRI; fluorouracil; 5-FU; leucovorin; irinotecan
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — veliparib; IFL protocol; Bevacizumab; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Veliparib + modified FOLFIRI ± bevacizumab (Experimental): Dosing of oral veliparib (200 mg) began 2 days prior to the start of FOLFIRI and continued twice a day (BID) for a total of 7 consecutive days. At the discretion of the Investigator, bevacizumab (5 mg/kg) could be administered intravenously (IV) immediately preceding FOLFIRI. Modified FOLFIRI was administered as irinotecan 180 mg/m^2 (90-minute infusion ± 30 minutes); leucovorin 400 mg/m^2 (90-minute infusion ± 30 minutes); and saline bolus (up to 15-minute infusion) immediately followed by fluorouracil 2400 mg/m^2 (46-hour continuous infusion ± 4 hours) starting on Day 1 of each 14-day cycle.
  Interventions: Drug: Veliparib; Drug: Modified FOLFIRI; Drug: Bevacizumab; Drug: Fluorouracil infusion
- Placebo + FOLFIRI ± bevacizumab (Placebo Comparator): Dosing of oral placebo (200 mg) began 2 days prior to the start of FOLFIRI and continued twice a day (BID) for a total of 7 consecutive days. At the discretion of the Investigator, bevacizumab (5 mg/kg) could be administered intravenously (IV) immediately preceding FOLFIRI. Standard FOLFIRI was administered as irinotecan 180 mg/m^2 (90-minute infusion ± 30 minutes); leucovorin 400 mg/m^2 (90-minute infusion ± 30 minutes); and fluorouracil bolus 400 mg/m^2 (up to 15-minute infusion) immediately followed by fluorouracil 2400 mg/m^2 (46-hour continuous infusion ± 4 hours) on Day 1 of each 14-day cycle.
  Interventions: Drug: Placebo; Drug: FOLFIRI; Drug: Bevacizumab; Drug: Fluorouracil infusion

INTERVENTIONS:
Drug: Veliparib — 200 mg oral dose beginning 2 days prior to the start of FOLFIRI and continuing twice a day (BID) for a total of 7 consecutive days
  Other Names: ABT-888
  Arms: Veliparib + modified FOLFIRI ± bevacizumab
Drug: Placebo — 200 mg oral dose beginning 2 days prior to the start of FOLFIRI and continuing twice a day (BID) for a total of 7 consecutive days
  Arms: Placebo + FOLFIRI ± bevacizumab
Drug: Modified FOLFIRI — Irinotecan 180 mg/m^2 (90-minute infusion ± 30 minutes); leucovorin 400 mg/m^2 (90-minute infusion ± 30 minutes); and saline bolus (up to 15-minute infusion) on Day 1 of each 14-day cycle
  Arms: Veliparib + modified FOLFIRI ± bevacizumab
Drug: FOLFIRI — Irinotecan 180 mg/m^2 (90-minute infusion ± 30 minutes); leucovorin 400 mg/m^2 (90-minute infusion ± 30 minutes); and fluorouracil bolus 400 mg/m^2 (up to 15-minute infusion) on Day 1 of each 14-day cycle
  Arms: Placebo + FOLFIRI ± bevacizumab
Drug: Bevacizumab — At the discretion of the Investigator, 5 mg/kg may be administered intravenously immediately preceding FOLFIRI dosing
  Other Names: Avastin
Drug: Fluorouracil infusion — 2400 mg/m^2 (46-hour continuous infusion ± 4 hours) starting on Day 1 of each 14-day cycle
  Other Names: 5-FU

SUMMARY:
This was a blinded, randomized, placebo-controlled Phase 2 multicenter study evaluating the efficacy and tolerability of veliparib plus irinotecan, fluorouracil, and leucovorin chemotherapy regimen (FOLFIRI) compared to placebo plus FOLFIRI in participants with previously untreated metastatic colorectal cancer. Participants could also have been treated with bevacizumab at the discretion of the Investigator.

DETAILED DESCRIPTION:
Participants were randomized to one of 2 groups: veliparib plus FOLFIRI ± bevacizumab (veliparib group) or placebo plus FOLFIRI ± bevacizumab (placebo group), and stratified by planned use of bevacizumab (planned bevacizumab use compared to unplanned use of bevacizumab) and regions of the world (North America versus rest of world). In this study, the term FOLFIRI was used to describe both the standard regimen containing a fluorouracil bolus that was administered to participants randomized to the placebo arm, and a modified regimen with a saline bolus that was administered to participants randomized to the veliparib arm. One cycle of protocol therapy consisted of 14 days, defined as Day -2 through Day 12. Dosing of oral veliparib/placebo began 2 days prior to the start of FOLFIRI and continued twice a day for a total of 7 consecutive days. At the discretion of the Investigator, bevacizumab could be administered intravenously immediately preceding FOLFIRI. Study visits were conducted on Day 1 and Day 8 of the first and second cycles, then on Day 1 of each subsequent cycle. Participants were to continue protocol therapy and study visits until they met one of the defined discontinuation criteria. When the Investigator determined that a participant met the criteria for discontinuation, a final visit was conducted. Participants were to have had one follow-up visit approximately 30 days after the last dose of protocol therapy. Sites began collecting post-treatment and survival information 4 weeks after the last clinical assessment. Post-baseline radiographic tumor assessment was to be conducted every 8 weeks from Cycle 1, Day 1 (prior to the start of a new cycle) until radiographic progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic adenocarcinoma of the colon or rectum
* At least 1 unresectable lesion on a CT (Computerized Tomography) scan that is measurable as defined by Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1
* ECOG (Eastern Cooperative Oncology Group) performance score of 0 or 1
* Adequate hematologic, renal and hepatic function

Exclusion Criteria:

* Prior anti-cancer treatment for metastatic colorectal cancer
* Prior exposure to PARP (poly ADP-ribose polymerase) inhibitors
* The last course of adjuvant or neoadjuvant chemotherapy must have ended > 12 months prior to Cycle 1 Day -2
* Any clinically significant and uncontrolled major medical condition
* Participant is pregnant or lactating
* Any medical condition, which in the opinion of the study Investigator, places the participant at an unacceptably high risk for toxicities
* For those receiving bevacizumab, standard medical exclusionary conditions apply

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All randomized participants. Although the study was terminated by the Sponsor, because all participants were evaluated for the primary end point, the study was considered to have Completed as planned.
Period: Overall Study
Arm/Group | Veliparib + Modified FOLFIRI ± Bevacizumab | Placebo + FOLFIRI ± Bevacizumab
Started | 65 | 65
Completed | 0 | 0
Not Completed | 65 | 65
Not completed — Death | 27 | 27
Not completed — Withdrew consent | 9 | 2
Not completed — Lost to Follow-up | 6 | 1
Not completed — Study Terminated by Sponsor | 21 | 34
Not completed — Other, not specified | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Veliparib + Modified FOLFIRI ± Bevacizumab | Placebo + FOLFIRI ± Bevacizumab | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (13.06) | 63.8 (9.04) | 61.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 44 | 40 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 62 | 64 | 126
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS): Time to Event
Description: PFS was defined as the number of days from the date the participant was randomized to the date the participant experienced an event of disease progression or death, whichever occurred first. All events of disease progression were included, whether the participant was still taking or had discontinued study drug. Events of death were included for participants who had not experienced an event of disease progression, if the death occurred within 8 weeks of the last evaluable disease progression assessment. If the participant did not have an event of disease progression and the participant had not died as defined above, data were censored at the date of the participant's last evaluable disease progression assessment. The PFS distribution was estimated using Kaplan-Meier methodology. Point estimates and 95% confidence intervals (95% CIs) for the PFS distribution quartiles are provided.
Time Frame: Every 8 weeks from Cycle 1, Day 1 until radiographic progression was observed. The maximum observed follow up duration at the progression-free survival analysis time was 579 days.
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Veliparib + Modified FOLFIRI ± Bevacizumab | Placebo + FOLFIRI ± Bevacizumab
Number analyzed (Participants) | 65 | 65
days
  25th Quartile | 221 [120 to 295] | 213 [121 to 233]
  50th Quartile | 361 [289 to 453] | 337 [233 to 421]
  75th Quartile | 534 [453 to NA] — The upper 95% CI limit was not estimable due to an insufficient number of participants with events, as indicated by NA. | 512 [421 to NA] — The upper 95% CI limit was not estimable due to an insufficient number of participants with events, as indicated by NA.
Statistical Analysis 1: Comparison: Veliparib + Modified FOLFIRI ± Bevacizumab vs Placebo + FOLFIRI ± Bevacizumab; Comparisons between treatment groups were performed using the Cox Proportional Hazard Model, stratified by planned bevacizumab use (planned use versus no planned use); Test type: Superiority; Hazard Ratio (HR) = 0.939, 95% CI 2-sided [0.596 to 1.480]

2. Secondary Outcome: Overall Survival (OS): Time to Event
Description: Overall survival was defined as the number of days from the date that the participant was randomized to the date of the participant's death. All events of death were included, regardless of whether the event occurred while the participant was still taking or had discontinued study drug. If a participant had not died, the data were censored at the date last known to be alive. The OS distribution was estimated using Kaplan-Meier methodology. Point estimates and 95% confidence intervals (95% CIs) for the OS distribution quartiles are provided.
Time Frame: Survival information was to be collected 4 wks after the last study visit, continuing every 4 wks for 1 yr, then every 8 wks for up to 2 more yrs or until death. The maximum observed follow up duration at the overall survival analysis time was 914 days.
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Veliparib + Modified FOLFIRI ± Bevacizumab | Placebo + FOLFIRI ± Bevacizumab
Number analyzed (Participants) | 65 | 65
days
  25th Quartile | 557 [391 to 616] | 512 [326 to 655]
  50th Quartile | 770 [609 to NA] — The upper 95% CI limit was not estimable due to an insufficient number of participants with events, as indicated by NA. | 811 [678 to NA] — The upper 95% CI limit was not estimable due to an insufficient number of participants with events, as indicated by NA.
  75th Quartile | NA [784 to NA] — NA= Not calculable due to insufficient survival events | NA [811 to NA] — NA= Not calculable due to insufficient survival events
Statistical Analysis 1: Comparison: Veliparib + Modified FOLFIRI ± Bevacizumab vs Placebo + FOLFIRI ± Bevacizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Hazard Ratio (HR) = 1.261, 95% CI 2-sided [0.738 to 2.156]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the proportion of participants with a complete (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1) for target lesions, assessed by computed tomography (CT). Complete response (CR) was defined as disappearance of all target lesions; partial response (PR) ≥30% decrease in the the sum of diameters of target lesions, taking as reference the baseline sum diameters. For participants who underwent surgery, ORR was not evaluated after surgery.
Time Frame: Per protocol, post-baseline tumor assessment was conducted every 8 weeks from Cycle 1 Day 1 until radiographic progression. The maximum observed follow up duration at the progression-free survival analysis time was 579 days.
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Veliparib + Modified FOLFIRI ± Bevacizumab | Placebo + FOLFIRI ± Bevacizumab
Number analyzed (Participants) | 65 | 65
Participants | 37 | 40
Statistical Analysis 1: Comparison: Veliparib + Modified FOLFIRI ± Bevacizumab vs Placebo + FOLFIRI ± Bevacizumab; Comparisons between treatment groups were performed using the Mantel-Haenszel method, stratified by planned bevacizumab use (planned use versus no planned use); Test type: Superiority; Mantel Haenszel; Difference in proportions = -4.62, 95% CI 2-sided [-21.4 to 12.1]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of veliparib/placebo administration until 30 days after the last dose of veliparib/placebo (up to 396 days).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of veliparib/placebo until 30 days after the last dose of veliparib/placebo and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Veliparib + Modified FOLFIRI ± Bevacizumab | Placebo + FOLFIRI ± Bevacizumab
All-Cause Mortality (participants affected / at risk) | 27/65 | 27/65
Serious Adverse Events (participants affected / at risk) | 30/65 | 33/65
Other Adverse Events (participants affected / at risk) | 59/65 | 60/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veliparib + Modified FOLFIRI ± Bevacizumab (N=65) | Placebo + FOLFIRI ± Bevacizumab (N=65)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 (5) | 3 (3)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 2 (2)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 1 (1)
TACHYARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 2 (3)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 9 (10) | 2 (2)
ENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 3 (5)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTRA-ABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
PROCTITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (2) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0)
EXTRAVASATION (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 0 (0)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 2 (2) | 0 (0)
HEPATOTOXICITY (Hepatobiliary disorders) | 1 (1) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1) | 1 (1)
CAMPYLOBACTER INFECTION (Infections and infestations) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1)
SERRATIA INFECTION (Infections and infestations) | 0 (0) | 1 (1)
STREPTOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (2)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (2) | 1 (1)
LACUNAR INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
DEVICE DISLOCATION (Product Issues) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (2) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veliparib + Modified FOLFIRI ± Bevacizumab (N=65) | Placebo + FOLFIRI ± Bevacizumab (N=65)
ANAEMIA (Blood and lymphatic system disorders) | 25 (59) | 12 (28)
LEUKOPENIA (Blood and lymphatic system disorders) | 11 (24) | 4 (8)
LYMPHOPENIA (Blood and lymphatic system disorders) | 4 (5) | 2 (3)
NEUTROPENIA (Blood and lymphatic system disorders) | 41 (108) | 23 (54)
ABDOMINAL PAIN (Gastrointestinal disorders) | 12 (16) | 22 (37)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (7) | 8 (9)
CONSTIPATION (Gastrointestinal disorders) | 9 (16) | 21 (29)
DIARRHOEA (Gastrointestinal disorders) | 29 (73) | 35 (103)
DRY MOUTH (Gastrointestinal disorders) | 4 (5) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 4 (4) | 2 (2)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 4 (5)
HAEMORRHOIDS (Gastrointestinal disorders) | 4 (5) | 4 (6)
NAUSEA (Gastrointestinal disorders) | 35 (69) | 40 (66)
STOMATITIS (Gastrointestinal disorders) | 15 (25) | 10 (14)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 4 (6)
VOMITING (Gastrointestinal disorders) | 26 (48) | 26 (38)
ASTHENIA (General disorders) | 16 (34) | 14 (41)
FATIGUE (General disorders) | 25 (38) | 24 (65)
MUCOSAL INFLAMMATION (General disorders) | 4 (7) | 14 (27)
OEDEMA PERIPHERAL (General disorders) | 5 (5) | 7 (7)
PYREXIA (General disorders) | 8 (15) | 11 (13)
BRONCHITIS (Infections and infestations) | 2 (7) | 5 (5)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (5) | 5 (5)
URINARY TRACT INFECTION (Infections and infestations) | 6 (8) | 4 (6)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (7) | 2 (2)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (3) | 4 (8)
WEIGHT DECREASED (Investigations) | 6 (6) | 5 (9)
DECREASED APPETITE (Metabolism and nutrition disorders) | 15 (21) | 19 (36)
DEHYDRATION (Metabolism and nutrition disorders) | 6 (9) | 6 (7)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 4 (5) | 9 (15)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 4 (9) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 10 (18) | 3 (3)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 4 (8) | 3 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (7)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (10) | 8 (11)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
DIZZINESS (Nervous system disorders) | 0 (0) | 4 (5)
DYSGEUSIA (Nervous system disorders) | 11 (11) | 6 (6)
HEADACHE (Nervous system disorders) | 10 (11) | 5 (12)
PARAESTHESIA (Nervous system disorders) | 5 (6) | 5 (6)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 3 (3) | 7 (7)
INSOMNIA (Psychiatric disorders) | 10 (10) | 8 (9)
DYSURIA (Renal and urinary disorders) | 5 (8) | 3 (3)
HAEMATURIA (Renal and urinary disorders) | 2 (2) | 5 (6)
PROTEINURIA (Renal and urinary disorders) | 3 (4) | 4 (6)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (8)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (9)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 17 (22)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 25 (28) | 18 (30)
DRY SKIN (Skin and subcutaneous tissue disorders) | 5 (12) | 3 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (8) | 4 (5)
HYPERTENSION (Vascular disorders) | 6 (12) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT02305758/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT02305758/SAP_001.pdf